CLINICAL TRIAL: NCT00347555
Title: Phase I, Double-Blinded, Placebo-Controlled Dosage-Escalation Study of the Safety and Immunogenicity of EBA-175 RII-NG Malaria Vaccine Administered Intramuscularly
Brief Title: Safety and Immunogenicity of EBA-175 RII-NG Malaria Vaccine Administered Intramuscularly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 04-059; N01AI80002C
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2012-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, falciparum, Plasmodium falciparum malaria, vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — aluminum phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group D (Experimental): 18 subjects 160 micrograms EBA-175+500 micrograms aluminum adjuvant; 2 subjects placebo.
  Interventions: Biological: Aluminum Phosphate; Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine
- Group A (Experimental): 18 subjects 5 micrograms EBA-175+500 micrograms aluminum adjuvant; 2 subjects placebo.
  Interventions: Biological: Aluminum Phosphate; Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine
- Group B (Experimental): 18 subjects 20 micrograms EBA-175+500 micrograms aluminum adjuvant; 2 subjects placebo.
  Interventions: Biological: Aluminum Phosphate; Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine
- Group C (Experimental): 18 subjects 80 micrograms EBA-175+500 micrograms aluminum adjuvant; 2 subjects placebo.
  Interventions: Biological: Aluminum Phosphate; Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine

INTERVENTIONS:
Biological: Aluminum Phosphate — 1.0 mg/mL (0.5 mg/0.5 mL per dose) aluminum as aluminum phosphate adjuvant; dosage 500 micrograms.
Drug: Placebo — 0.5 mL normal saline placebo. Sodium phosphate buffer (10 mM sodium phosphate and 150 mM sodium chloride).
Biological: EBA-175 RII-NG Malaria Vaccine — White, translucent, cloudy, nonparticulate liquid suspension. Recombinant Plasmodium falciparum erythrocyte-binding antigen 175 kDa Region II-nonglycosylated (EBA-175 RII-NG) absorbed to aluminum phosphate adjuvant; dosage levels 5, 20, 80, and 160 micrograms.

SUMMARY:
Malaria is an illness caused by a parasite (an animal or plant that lives in or on a host) that enters the human body through the bite of an infected mosquito. The purpose of this study is to find out about the safety of an experimental malaria vaccine and whether the vaccine causes humans to produce antibodies (proteins made by the body's immune system to help control or prevent infection). Four strengths of the vaccine will be tested. The lowest strength of the vaccine will be tested before the next higher strength is tested. Each dosage (shot) of vaccine will be given to 18 people in 4 dosage groups on Day 0, at 1 month and at 6 months. Two people in each dosage group will receive injections of a placebo (contains no medication). Participants will include 80 healthy adults between 18 and 40 years of age. Multiple blood draws will occur over the duration of the study. Participants will be involved in study related procedures for approximately 13 months.

DETAILED DESCRIPTION:
This study is a phase I, double-blinded, placebo-controlled, dosage-escalation study of the safety and immunogenicity of EBA-175 RII-NG malaria vaccine administered intramuscularly. The vaccine is a recombinant Plasmodium falciparum (Pf) erythrocyte-binding antigen 175 kDa Region II-nonglycosylated (EBA-175 RII-NG) adsorbed to aluminum phosphate adjuvant. The study is being conducted at Baylor College of Medicine, Houston, Texas. Eighty healthy subjects, between the ages of 18 and 40 years, males and females, will be recruited from Houston, Texas, and will participate in the study for approximately 13 months. Subjects will be randomized to receive 3 doses of the vaccine or saline placebo by the intramuscular route in a 9:1 ratio at 0, 1 and 6 months. The safety and immunogenicity of ascending dosages of the vaccine will be assessed. Eighteen subjects will receive vaccine at each of the following dosage levels: 5, 20, 80 and 160 micrograms. Two subjects will receive placebo for each dosage level. Dosage escalation will proceed only after review of the 2-week safety data of the 2 initial doses of the prior dosage level. The primary study objective is to assess the safety and reactogenicity (tolerability) of ascending dosages of EBA-175 RII-NG vaccine among healthy subjects given in 3 intramuscular doses at 0, 1 and 6 months. The secondary study objective is to evaluate the immunogenicity of the EBA-175 RII-NG vaccine by measuring anti-EBA-175 RII-NG antibodies using enzyme-linked immunosorbent assay (ELISA), anti-parasite antibodies by indirect fluorescence antibody test (IFAT), inhibition of binding of EBA-175 RII-NG to red blood cells (RBCs), and inhibition of Pf growth in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and healthy nonpregnant females between the ages of 18 and 40 years.
* Females of childbearing potential must agree to practice adequate contraception for the entire study period (including abstinence; hormonal contraception; condoms with spermicidal agents; surgical sterilization; or vasectomized partner).
* Good health as determined by screening medical history, physical examination, and routine laboratory assessments.
* Willingness to comply with protocol requirements.
* Ability to provide informed consent before any protocol procedures are performed.
* Availability for follow up for 12 months after the first immunization dose.

Exclusion Criteria:

* Regular use of medications other than vitamins and contraceptives.
* Current or recent (within the last 4 weeks) treatment with parenteral, inhaled, or oral corticosteroids (intranasal steroids are acceptable), or other immunosuppressive agents, or chemotherapy.
* History of splenectomy.
* Abnormal screening laboratory values. Any abnormal screening value for any screening test, except reticulocyte count (even if in subsequent tests the value is within normal range) will exclude the subject from the study. An exception to this rule is the glucose measurement. Random plasma glucose will be measured on all subjects during the screening visit. Values higher than 109 mg/dl will be confirmed by a repeat fasting glucose measurement.
* History of or current medical, occupational, social or family problems as a result of alcohol or illicit drug use.
* History of moderate to severe mental illness, as defined by symptoms interfering with social or occupational function or suicidal thoughts/attempts.
* History of receiving blood or blood products (such as blood transfusion, platelet transfusion, immunoglobulins, hyperimmune serum) in the previous 6 months.
* Vaccination with a live vaccine within the past 30 days or with a nonreplicating, inactivated, or subunit vaccine within the last 14 days.
* Known hypersensitivity to components of the vaccine (EBA-175 RII-NG, sucrose, or aluminum adjuvant).
* History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic and autoimmune/inflammatory conditions.
* History of anaphylaxis or severe hypersensitivity reaction.
* Severe asthma, as defined by an emergency room visit or hospitalization within the last 12 months.
* Pregnant or breastfeeding women, or women unwilling to use effective contraception during the study period.
* Acute illness, including temperature >100 degrees F within one week of vaccination.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days.
* Identification of any condition that, in the opinion of the investigator, would affect the ability of the subject to understand or comply with the study protocol or would jeopardize the safety or rights of a subject participating in the study.
* History of malignancy, including hematologic and skin cancers, or known immunodeficiency syndrome.
* History of malaria infection or receipt of a malaria vaccine.
* History of travel to malaria-endemic area or receipt of antimalarial prophylaxis in the past 12 months.
* Planned travel to a malaria-endemic area during the course of the study.
* Pre-medication with analgesic or antipyretic in the 6 hours prior to vaccination, or planned medication with analgesic or antipyretic in the 24 hours following vaccination. This should not preclude subjects receiving such medication if the need arises.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of injection site and systemic adverse events (AEs). | Duration of study.

SECONDARY OUTCOMES:
Relative binding inhibition of recombinant EBA-175 RII-NG to human RBCs in vitro in the presence of serum from immunized individuals. | Days 0, 14, 28, 42, 180, and 194.
Anti-parasite antibodies by indirect fluorescence antibody test (IFAT). | Days 0, 14, 28, 42, 180, and 194.
Anti-EBA-175 RII-NG antibody level by ELISA. | Days 0, 14, 28, 42, 180, and 194.
Relative growth inhibition of Pf in human RBCs cultured in vitro in the presence of serum from immunized individuals. | Days 0, 14, 28, 42, 180, and 194.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States